CLINICAL TRIAL: NCT01121341
Title: ESOS (Endoscopic Saphenous Harvesting With an Open CO2 System) Trial: a Prospective Randomized Trial for Coronary Artery Bypass Grafting (CABG) Surgery.
Brief Title: ESOS (Endoscopic Saphenous Harvesting With an Open CO2 System) Trial
Acronym: ESOS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Collaborators: LivaNova (Industry)
Responsible Party: Silvana Barbaro and Serenella Scipioni, Azienda Ospedaliera San Giovanni Battista
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEI/7
Record Dates: First submitted 2010-05-07; First posted 2010-05-12 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2010-04

CONDITIONS: Coronary Artery Bypass Grafting Surgery
Keywords: Endoscopic vein harvesting; Saphenous vein; Conventional vein harvesting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVOH (Experimental): Procedure: Endoscopic vein with an open CO2 system harvesting
  Interventions: Procedure: Vein harvesting
- OVH (Active Comparator): Procedure: Conventional vein harvesting
  Interventions: Procedure: Vein harvesting

INTERVENTIONS:
Procedure: Vein harvesting — Endoscopic versus conventional vein harvesting

SUMMARY:
The ESOS (Endoscopic Saphenous harvesting with an Open CO2 System) trial is a prospective randomized trial for coronary artery bypass grafting (CABG) surgery to compare endoscopic open CO2 harvesting system versus conventional vein harvesting.

DETAILED DESCRIPTION:
The ESOS (Endoscopic Saphenous harvesting with an Open CO2 System) trial is a prospective randomized trial for coronary artery bypass grafting (CABG) surgery to compare and to test improvement in wound healing, quality of life, safety/efficacy, cost-effectiveness, short and long-term outcomes and vein-graft patency after endoscopic open CO2 harvesting system versus conventional vein harvesting.

ELIGIBILITY:
Inclusion Criteria:

* Elective planned CABG surgery
* First isolated CABG surgery

Exclusion Criteria:

* Emergency revascularization: patients with hemodynamic instability or requiring inotropic or intra-aortic balloon support
* Previous cardiac surgery
* Planned concomitant valve surgery
* Very varicous veins
* Previous saphenectomy
* History of deep vein thrombosis
* History of suffered trauma on the lower extremity
* Preoperative legs immobilization
* Previous leg wound complications
* Coexisting illness with life expectancy < five years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Morbidity hypothesis | six weeks
  When compared to Conventional vein-graft harvesting (CVH) in CABG surgery
  · Does Endoscopic vein-graft open CO2 system harvesting (EVOH) reduce postoperative wound complications (composite endpoint of all complications or individual complications) assessed with ASEPSIS score?
Patient satisfaction hypothesis | six weeks
  · Does EVOH improve patient satisfaction, postoperative leg pain and quality of life assessed with VAS score and EUROQol-5D?
  * To compare health-related quality of life for the two treatment arms (EVOH/CVH) by intention-to-treat
  * To identify factors in addition to treatment assignment that are associated with variations in quality of life outcomes
Resource utilization hypothesis | six weeks
  When compared to Conventional vein-graft harvesting (CVH) in CABG surgery
  · Does EVOH affect resource utilization?
  * Harvesting time related to the length of vein segments
  * Harvesting closure time
  * CABG time
  * Mobility time
  * Hospital length of stay
  * Re-exploration for bleeding due to vein-graft bleed
  * Readmission for leg wound complications
  * Need for outpatient wound management resources
  * To compare total medical costs for the two treatment arms (EVOH/CVH) by intention-to-treat
Quality of vein harvesting hypothesis | six weeks
  When compared to Conventional vein-graft harvesting (CVH) in CABG surgery
  * Do EVOH compromises the quality of venous conduit harvested?
    * Number of harvested veins requiring repair
    * Number of repairs to each vein
    * Re-exploration for bleeding due to vein-graft bleed
    * Histological integrity
  * Specific secondary subanalysis adjusted for:
    * Preparation solution of the vein conduit
      * 20 ml autologous blood
      * 0,5 ml heparin (5000UI/ml) = 2500 UI
      * 2 ml papavarine (30mg/ml) = 60 mg
    * Uncontrolled distension pressure/ no touch technique harvesting

SECONDARY OUTCOMES:
Vein-graft patency hypothesis | six weeks
  Does EVH Open-CO2 system influence and improve vein-graft patency?
  * Assessment of systemic carbon dioxide absorption with respiratory and hemodynamic parameters
  * Assessment of vein-graft patency with:
    * vein conduit quality [diameter/well thickness]
    * vein segments above/below the knee
    * target coronary artery grafted territory
    * target coronary artery diameter
    * target coronary artery stenosis
    * target coronary artery severity disease
    * ascending aorta disease
    * composite /uncomposite graft
    * left ventricular function
outcome hypothesis | 18 months
  § Detection of long-term outcomes:
  * MACE (major adverse cardiac events): death; myocardial infarction; revascularization (PCI or CABG) for ischemia or angina recurrence
  * MACE related to vein-graft failure
  * GF (vein-graft failure): at least 75% of stenosis;
  * GO (vein-graft occlusion) at angiographic study
  * to identify factors in addition to treatment assignment that are associated with variations in long-term outcomes and graft patency
  * baseline demographic characteristics and medications used of two treatment arms (EVOH/CVH)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Campanella, MD, Study Chair — Department of Thoracic and Cardiovascular Surgery, San Giovanni Battista of Turin Hospital, Corso Bramante 88/90, 10126 Turin, Italy; Mauro Rinaldi, MD, PhD, Principal Investigator — Department of Thoracic and Cardiovascular Surgery, San Giovanni Battista of Turin Hospital, Corso Bramante 88/90, 10126 Turin, Italy
Locations (1):
- Azienda Ospedaliero-Universitaria San Giovanni Battista di Torino, Turin, Piedmont, Italy

REFERENCES:
- [Derived] Campanella A, Bergamasco L, Macri L, Asioli S, Devotini R, Scipioni S, Barbaro S, Rispoli P, Rinaldi M. Endoscopic Saphenous harvesting with an Open CO2 System (ESOS) trial for coronary artery bypass grafting surgery: study protocol for a randomized controlled trial. Trials. 2011 Nov 18;12:243. doi: 10.1186/1745-6215-12-243. PMID 22098690